CLINICAL TRIAL: NCT04365803
Title: Comparison Between Histological VABB and Histological Post-surgery in Patient With Complete Pathological Response After Neoadjuvant Systemic Treatment: Pilot Study
Brief Title: Histology VABB-Histology Post Surgery Pilot Project (BETTY Trial)
Acronym: BETTY
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: IEO 0758/
Record Dates: First submitted 2020-04-24; First posted 2020-04-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer
Keywords: breast cancer; vacuum assisted breast biopsy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient with radiological complete response: patient with radiological complete response after neoadjuvant chemotherapy
  Interventions: Procedure: vacuum-assisted breast biopsy

INTERVENTIONS:
Procedure: vacuum-assisted breast biopsy — patient with radiological complete response after neoadjuvant chemotherapy undergo to vacuum assisted breast biopsy and the to definitive surgery

SUMMARY:
Pilot study on patients with invasive ductal breast cancer triple negative or receptor tyrosine-protein kinase erbB-2 (HER2) overexpressed, any axillary lymphnodes status (any cN), candidates to neoadjuvant chemotherapy.

The principal endpoint of the study will be the accuracy of the result of the histological examination of the Vacuum- Assisted Breast Biopsy (VABB) performed pre-surgery in comparison to the result of the histological examination of the definitive surgical intervention in patients with radiological complete response at Magnetic resonance imaging (MRI) done after the end of neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
The study articulates in five phases:

Phase one: acquisition of the informed consent followed by positioning a clip into the cancer bed (by radiologist) if not already present; Phase two: after radiological confirmation of pathological Complete Response (pCR) done performing breast ultrasound, MRI and 18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose positron emission tomography (18-FDG-PET) after neoadjuvant chemotherapy the patient becomes candidate to VABB pre surgery.

Phase three: the patient has VABB within 15 day from the term of neoadjuvant chemotherapy Phase four: definitive surgical intervention within 30 days from the end of the neoadjuvant chemotherapy Phase five: verification of correspondence between histology of VABB and definitive histology.

The study hypothesis is that VABB could be used in the patients with pCR to the imaging post-neoadjuvant chemotherapy to confirm sensibility and specificity of 18 FDG TC PET and breast MRI to show the absence of breast cancer.

The use of VABB with negative histology result could bring to a therapeutic gold standard without over surgical treatment

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 aa;
* histological diagnosis done at European Institute of Oncology (if not, to does revision of pathological material);
* invasive ductal breast cancer triple negative or HER2 overexpressed, any cN;
* neoadjuvant standard systemic treatment after surgery +/- trastuzumab;
* propose of conservative or demolitive surgery;
* M0
* cancer bed identified pre neoadjuvant chemotherapy by clip

Exclusion Criteria:

* multicentric or bilateral breast cancer
* mammography microcalcifications
* in situ breast carcinoma
* positive anamnesis for previous breast cancer
* positive anamnesis for medical or psychological conditions that prevent membership study

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with triple negative or HER2 over-expressed breast cancer with radiological complete response after neoadjuvant chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 22 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the accuracy of histological examination of the VABB performed pre-surgery | 45 days
  Identification of percentage of cases with correspondence between histology of VABB presurgery and histology of definitive surgery in patients with complete radiological response after neoadjuvant chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Elisabetta Rossi, MD, Principal Investigator — European Institute of Oncology
Locations (1):
- European Instituto of Oncology, Milan, Italy